CLINICAL TRIAL: NCT01236001
Title: Multi-center, Observational, Drug-utilization Study in Belgium to Evaluate the Use of VIMPAT® in Clinical Practice as Adjunctive Treatment of Partial Onset Epilepsy in Subjects Aged 16 and Older.
Brief Title: Belgian Drug-utilization Study to Evaluate the Use of VIMPAT® as Adjunctive Treatment of Partial Onset Seizures in Subjects Aged 16 and Older
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: SP1021
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Results first posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Seizures
Keywords: Lacosamide; Vimpat®
MeSH Terms: conditions — Seizures | interventions — Lacosamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vimpat® treatment: Patients who started VIMPAT® treatment before enrollment and patients who started VIMPAT® on/after enrollment.
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide
  Other Names: VIMPAT®

SUMMARY:
Observational study at the request of the Belgian Institut National d'Assurance Maladie-Invalidité / Rijksinstituut voor Ziekte-en Invaliditeits Verzekering INAMI/RIZIV:

* type of patient treated with VIMPAT®
* VIMPAT® dose
* Effect of VIMPAT® on evolution of seizure control
* Persistence rate at 6 months in terms of treatment duration
* Discontinuation rate
* Description of any changes in other epilepsy therapies
* Safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent form
* Subject/legal representative is considered reliable and capable of adhering to the medication intake according to the judgement of the investigator
* Based on the investigators clinical judgement, the subjects' seizure activity is uncontrolled on current therapy and it is in the subjects' best interest to be prescribed an antiepileptic drug (AED) as adjunctive therapy. The choice to prescribe VIMPAT® as adjunctive therapy is made by the treating investigator
* The subject is aged 16 or older
* The subject has a diagnosis of epilepsy with partial-onset seizures according to the label
* The subject has a medication history with at least 3 AED therapies (lifetime and/or concomitant) with treatment failure: due to insufficient efficacy, due to significant adverse events
* Sufficient data on the clinical situation before start of VIMPAT® and information on VIMPAT® dosing are present in the subject's medical record for patients on treatment with VIMPAT® at the time of enrollment into the study

Exclusion Criteria:

* The subject has previously participated in this study or has participated in a clinical trial within the last 2 months
* The subject has a history of chronic alcohol or drug abuse within the last 6 months
* The subject has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the subject's ability to participate in this study
* The subject has a known hypersensitivity and/or allergy to soya, peanuts, or any component of VIMPAT®
* The subject is pregnant or lactating
* The subject has a known AV-block degree 2 or 3
* The subject is expected to be insufficiently compliant with contraception.
* The subject has a history of suicide attempt, has received professional counseling for suicidal ideation, or is currently experiencing active suicidal ideation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Routine clinical practice of neurologist / neuropsychiatrist / neurosurgeon / neuropediatrician Sampling based upon request by the Belgian reimbursement authorities: request to report on 100 patients
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (17):
- Belgium (17):
  - Aalst
  - Antwerp
  - Assebroek
  - Bruges
  - Brussels
  - Charleroi
  - Duffel
  - Ghent
  - Hasselt
  - La Louvière
  - Leuven
  - Liège
  - Marche-en-Famenne
  - Mons
  - Montegnée - Liege
  - Ottignies-Louvain-la-Neuve
  - Yvoir

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational study began enrollment in September 2010. The last patient visit occurred in March 2012. There were 22 study sites in Belgium.
Pre-assignment Details: The Safety Set (SS) and Full Analysis Set (FAS) both consisted of 192 subjects. The SS consisted of all enrolled subjects who received at least one dose of VIMPAT (before or during the study). The FAS consists of all enrolled subjects.
Groups:
- Patients Treated With VIMPAT® Prior to Enrollment: Patients who started VIMPAT® treatment before enrollment.
- Patients Who Started VIMPAT® Treatment on/After Enrollment: Patients who started VIMPAT® treatment on/after enrollment.
Period: Overall Study
Arm/Group | Patients Treated With VIMPAT® Prior to Enrollment | Patients Who Started VIMPAT® Treatment on/After Enrollment
Started | 105 | 87
Completed | 87 | 65
Not Completed | 18 | 22
Not completed — Adverse Event | 5 | 14
Not completed — Lack of Efficacy | 6 | 6
Not completed — Lost to Follow-up | 6 | 1
Not completed — Incompliance | 1 | 0
Not completed — Planned Visit After End of Study | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Set (SS) consists of all enrolled subjects who received at least one dose of VIMPAT® (before or during the study).
  The SS was used to analyze demographic data and baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Treated With VIMPAT® Prior to Enrollment | Patients Who Started VIMPAT® Treatment on/After Enrollment | Total
Number analyzed (Participants) | 105 | 87 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 4
  Between 18 and 65 years | 97 | 81 | 178
  >=65 years | 5 | 5 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 40.1 (13.4) | 43.3 (14.0) | 41.5 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 52 | 112
  Male | 45 | 35 | 80
Region of Enrollment [Number; unit: participants]
  Belgium | 105 | 87 | 192

OUTCOME MEASURES:

1. Primary Outcome: Mean Total Daily Dose of VIMPAT® (mg) at Baseline
Description: Mean total daily dose at baseline will be only provided for subjects who were already treated by VIMPAT® at Baseline.
Time Frame: Baseline
Population: Of the 192 subjects in the Safety Set (SS), 105 subjects were treated with Vimpat at Baseline are included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/day of Vimpat
Arm/Group | Patients Treated With VIMPAT® Prior to Enrollment
Number analyzed (Participants) | 105
mg/day of Vimpat | 272.1 (114.4)

2. Primary Outcome: Mean Total Daily Dose of VIMPAT® (mg) at 3 Months
Time Frame: 3 months
Population: Of the 192 subjects in the Safety Set (SS), 137 subjects had Vimpat daily dosing information available at the 3-month visit and are included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/day of Vimpat
Groups:
- Total Population: Patients who started VIMPAT® treatment before enrollment and patients who started VIMPAT® on/after enrollment.
Arm/Group | Patients Treated With VIMPAT® Prior to Enrollment | Patients Who Started VIMPAT® Treatment on/After Enrollment | Total Population
Number analyzed (Participants) | 74 | 63 | 137
mg/day of Vimpat | 316.2 (106.7) | 211.1 (77.4) | 267.9 (107.7)

3. Primary Outcome: Mean Total Daily Dose of VIMPAT® (mg) at 6 Months
Time Frame: 6 months
Population: Of the 192 subjects in the Safety Set (SS), 154 subjects had Vimpat dosing data available at the 6-month visit and are included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/day of Vimpat
Arm/Group | Patients Treated With VIMPAT® Prior to Enrollment | Patients Who Started VIMPAT® Treatment on/After Enrollment | Total Population
Number analyzed (Participants) | 87 | 67 | 154
mg/day of Vimpat | 329.9 (119.5) | 262.7 (103.9) | 300.6 (117.5)

4. Primary Outcome: Galenic Formulation Repartition in Subjects Treated by VIMPAT® at Baseline
Description: This outcome will be only provided for subjects who were already treated by VIMPAT® at Baseline.
  VIMPAT is available as tablet and oral solution formulation in Belgium. The use of each galenic formulation will be presented with number of subjects by formulation.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Patients Treated With VIMPAT® Prior to Enrollment
Number analyzed (Participants) | 105
participants
  Tablet | 104
  Oral Solution | 1

5. Primary Outcome: Galenic Formulation Repartition in Subjects Treated by VIMPAT® at 3 Months
Description: VIMPAT is available as tablet and oral solution formulation in Belgium. The use of each galenic formulation will be presented with number of subjects by formulation.
Time Frame: 3 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Patients Treated With VIMPAT® Prior to Enrollment | Patients Who Started VIMPAT® Treatment on/After Enrollment | Total Population
Number analyzed (Participants) | 74 | 63 | 137
participants
  Tablet | 74 | 63 | 137
  Oral Solution | 0 | 0 | 0

6. Primary Outcome: Galenic Formulation Repartition in Subjects Treated by VIMPAT® at 6 Months
Description: as for outcome 5
Time Frame: 6 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Patients Treated With VIMPAT® Prior to Enrollment | Patients Who Started VIMPAT® Treatment on/After Enrollment | Total Population
Number analyzed (Participants) | 87 | 67 | 154
participants
  Tablet | 87 | 67 | 154
  Oral Solution | 0 | 0 | 0

7. Secondary Outcome: Percentage of Subjects Who Received Concomitant Antiepileptic Drug Treatment
Description: Concomitant antiepileptic drug (AED) treatments are defined as treatments which started after or at the date of the first administration of VIMPAT®.
Time Frame: From baseline to study termination (6 months)
Population: Of the 192 subjects in the Safety Set (SS), 192 are included in this analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Patients Treated With VIMPAT® Prior to Enrollment | Patients Who Started VIMPAT® Treatment on/After Enrollment | Total Population
Number analyzed (Participants) | 105 | 87 | 192
percentage of patients | 98.1 | 96.6 | 97.4

8. Secondary Outcome: Treatment Persistence of VIMPAT® After 6 Months
Description: Treatment persistence is defined as the percentage of subjects being treated under VIMPAT® after a given duration (>=6 months).
Time Frame: >=6 months
Population: Of the 192 subjects in the Safety Set (SS), 192 are included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Patients Treated With VIMPAT® Prior to Enrollment | Patients Who Started VIMPAT® Treatment on/After Enrollment | Total Population
Number analyzed (Participants) | 105 | 87 | 192
percentage of participants | 95.2 | 56.3 | 77.6

9. Secondary Outcome: Percentage of Subjects by Category of Clinical Evolution of Seizure Control at Baseline
Description: This outcome will be only provided for subjects who were already treated by VIMPAT® at Baseline.
  Clinical evolution of seizures following administration of VIMPAT compared to baseline before start of VIMPAT. The evolution of seizure control is subjectively assessed by the investigator on a four categorical scale, with options being 1=worsened, 2=stable, 3=improved, 4=much improved. If seizure control is worse, the investigator will try to document the reason.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Patients Treated With VIMPAT® Prior to Enrollment
Number analyzed (Participants) | 105
percentage of participants
  Much Improved | 16.2
  Improved | 39.0
  Stable | 30.5
  Worsened | 2.9
  Unknown | 11.4

10. Secondary Outcome: Percentage of Subjects by Category of Clinical Evolution of Seizure Control at 3 Months
Description: Clinical evolution of seizures following administration of VIMPAT compared to baseline before start of VIMPAT. The evolution of seizure control is subjectively assessed by the investigator on a four categorical scale, with options being 1=worsened, 2=stable, 3=improved, 4=much improved. If seizure control is worse, the investigator will try to document the reason.
Time Frame: 3 months
Population: Of the 192 subjects in the Safety Set (SS), 152 subjects had Vimpat daily dosing information available at the 3-month visit and are included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Patients Treated With VIMPAT® Prior to Enrollment | Patients Who Started VIMPAT® Treatment on/After Enrollment | Total Population
Number analyzed (Participants) | 78 | 74 | 152
percentage of participants
  Much improved | 16.7 | 16.2 | 16.4
  Improved | 43.6 | 33.8 | 38.8
  Stable | 34.6 | 35.1 | 34.9
  Worsened | 5.1 | 9.5 | 7.2
  Unknown | 0 | 5.4 | 2.7

11. Secondary Outcome: Percentage of Subjects by Category of Clinical Evolution of Seizure Control at 6 Months
Description: as for outcome 10
Time Frame: 6 months
Population: Of the 192 subjects in the Safety Set (SS), 168 subjects had Vimpat dosing data available at the 6-month visit and are included in this analysis.
Measure: Number; unit: percentage of participants
Groups:
- Total Population: Patients who started VIMPAT® treatment before enrollment and patients who started VIMPAT® treatment on/after enrollment.
Arm/Group | Patients Treated With VIMPAT® Prior to Enrollment | Patients Who Started VIMPAT® Treatment on/After Enrollment | Total Population
Number analyzed (Participants) | 95 | 73 | 168
percentage of participants
  Much improved | 18.9 | 19.2 | 19.0
  Improved | 35.8 | 38.4 | 36.9
  Stable | 40.0 | 34.2 | 37.5
  Worsened | 5.3 | 8.2 | 6.5

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected during the course of the trial, which was approximately 2 years.
Description: Adverse Events refer to the Safety Set (SS). The Safety Set (SS) consisted of all subjects who were randomized and received at least 1 dose of study medication.
Groups:
- Vimpat® Treatment: Reported Adverse Events is a combination of both patients who started VIMPAT® treatment before enrollment and patients who started VIMPAT® treatment on/after enrollment.
Arm/Group | Vimpat® Treatment
Serious Adverse Events (participants affected / at risk) | 8/192
Other Adverse Events (participants affected / at risk) | 74/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vimpat® Treatment (N=192)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Meningitis herpes (Infections and infestations) | 1 (1)
Status epilepticus (Nervous system disorders) | 3 (3)
Convulsion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vimpat® Treatment (N=192)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 5 (5)
Diplopia (Eye disorders) | 5 (5)
Dry eye (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (9)
Constipation (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 14 (14)
Gait disturbance (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 19 (19)
Somnolence (Nervous system disorders) | 9 (9)
Headache (Nervous system disorders) | 7 (7)
Ataxia (Nervous system disorders) | 4 (4)
Disturbance in attention (Nervous system disorders) | 3 (3)
Cognitive disorder (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Dysarthria (Nervous system disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Confusional state (Psychiatric disorders) | 4 (4)
Depressed mood (Psychiatric disorders) | 3 (3)
Abnormal dreams (Psychiatric disorders) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2)
Depressive symptom (Psychiatric disorders) | 2 (2)
Acute stress disorder (Psychiatric disorders) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1)
Conduct disorder (Psychiatric disorders) | 1 (1)
Decreased interest (Psychiatric disorders) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1)
Middle insomnia (Psychiatric disorders) | 1 (1)
Obsessive-compulsive disorder (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Sleep walking (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.